CLINICAL TRIAL: NCT00927082
Title: A Follow-up Study to Evaluate the Long-term Post Treatment Effects of Peginterferon Alfa-2a (PEG-IFN) in Patients With HBeAg Positive Chronic Hepatitis B From the Original Study WV19432(NEPTUNE).
Brief Title: A Follow-Up Study to WV19432, to Evaluate Long Term Post-Treatment Effects of PEGASYS (Peginterferon Alfa-2a(40KD))in Patients With HBeAg Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MV22430
Record Dates: First submitted 2009-06-16; First posted 2009-06-24 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (4):
- PEG-IFN 90mcg 24 Wks (Experimental): Participants received Pegasys (Pegylated interferon alfa-2a [PEG-IFN]) 90 micrograms (mcg) subcutaneously (SC) once a week for 24 weeks in Study WV19432 and entered follow-up (FU) Study MV22430.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- PEG-IFN 180mcg 24 Wks (Experimental): Participants received PEG-IFN 180 mcg SC once a week for 24 weeks in Study WV19432 and entered FU Study MV22430.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- PEG-IFN 90mcg 48 Wks (Experimental): Participants received PEG-IFN 90 mcg SC once a week for 48 weeks in Study WV19432 and entered FU Study MV22430.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- PEG-IFN 180mcg 48 Wks (Experimental): Participants received PEG-IFN 180 mcg SC once a week for 48 weeks in Study WV19432 and entered FU Study MV22430.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 90 or 180 micrograms/week sc for 24 or 48 weeks in original study (WV19432). No study treatment in long-term post-treatment follow-up study (MV22430)

SUMMARY:
This study is a long-term post-treatment follow-up to study WV19432, which evaluated the efficacy and safety of PEGASYS in patients with HBeAg positive chronic hepatitis B (CHB).Patients who received treatment with PEGASYS, and completed follow-up, are eligible to enter this post-treatment follow-up study. The anticipated time on study was 5 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for Study WV19432
* Patients who have completed treatment and follow-up on study WV19432

Exclusion Criteria:

* As for Study WV19432

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2009-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Fitzroy, Victoria, Australia
- Brazil (5):
  - Salvador, Estado de Bahia
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
- China (4):
  - Beijing
  - Changsha
  - Guangzhou
  - Shanghai
- Hong Kong, Hong Kong
- New Zealand (2):
  - Auckland
  - Hamilton
- Russia (3):
  - Saint Petersburg
  - Samara
  - Stavropol
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Songkhla

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 10 April 2009 to 05 November 2014. A total of 383 participants were recruited from 31 centers across 9 countries (Australia, New Zealand, China, Taiwan, Singapore, Korea, Thailand, Brazil, and Russia).
Period: Overall Study
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Started | 91 | 87 | 108 | 97
Completed | 79 | 77 | 86 | 78
Not Completed | 12 | 10 | 22 | 19
Not completed — Lost to Follow-up | 9 | 8 | 12 | 16
Not completed — Withdrawal by Subject | 3 | 2 | 7 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Screen fail,Participant migrated,Unknown | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat analysis population included all participants who had received at least one dose of study medication in study WV19432 and provided informed consent for study MV22430. Participants were analyzed according to the treatment groups to which they had been randomized.
Groups:
- PEG-IFN 90mcg 24 Wks: Participants received PEG-IFN 90 mcg SC once a week for 24 weeks in Study WV19432 and entered FU Study MV22430.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks | Total
Number analyzed (Participants) | 91 | 87 | 108 | 97 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.73) | 34.5 (10.54) | 34.3 (10.82) | 34.2 (10.78) | 33.9 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 23 | 33 | 35 | 125
  Male | 57 | 64 | 75 | 62 | 258

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Envelope Antigen (HBeAg) Seroconversion.
Description: HBeAg seroconversion was defined as the absence of HBeAg (a negative result for HBeAg) and the presence of anti-HBe (a positive result for anti-HBe). Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: The Per Protocol (PP) population included participants who satisfied key inclusion/exclusion criteria of Study WV19432, received at least 4 doses of PEG-IFN, and provided informed consent for Study MV22430. Analysis was performed per the treatment received and not the randomized treatment. Four participants switched treatment groups for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  End of Treatment (EOT) | 9.7 [4.5 to 17.6] | 14.6 [8.0 to 23.7] | 19.8 [12.7 to 28.7] | 31.6 [22.4 to 41.9]
  FU Year 1 | 20.4 [12.8 to 30.1] | 31.5 [22.0 to 42.2] | 27.4 [19.1 to 36.9] | 35.8 [26.2 to 46.3]
  FU Year 2 | 26.9 [18.2 to 37.1] | 37.1 [27.1 to 48.0] | 30.2 [21.7 to 39.9] | 47.4 [37.0 to 57.9]
  FU Year 3 | 38.7 [28.8 to 49.4] | 40.4 [30.2 to 51.4] | 34.0 [25.0 to 43.8] | 52.6 [42.1 to 63.0]
  FU Year 4 | 37.6 [27.8 to 48.3] | 44.9 [34.4 to 55.9] | 41.5 [32.0 to 51.5] | 49.5 [39.1 to 59.9]
  FU Year 5 | 41.9 [31.8 to 52.6] | 44.9 [34.4 to 55.9] | 40.6 [31.1 to 50.5] | 48.4 [38.0 to 58.9]

2. Secondary Outcome: Percentage of Participants With HBeAg Loss.
Description: HBeAg loss is defined as the absence of HBeAg (i.e. a negative result for HBeAg). Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: The PP population included participants who satisfied key inclusion and exclusion criteria of study WV19432, received at least 4 doses of PEG-IFN, and provided informed consent for study MV22430. Analysis was performed as per the treatment received and not the randomized treatment. Four participants switched treatment groups for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 9.7 [4.5 to 17.6] | 14.6 [8.0 to 23.7] | 19.8 [12.7 to 28.7] | 33.7 [24.3 to 44.1]
  FU Year 1 | 23.7 [15.5 to 33.6] | 31.5 [22.0 to 42.2] | 30.2 [21.7 to 39.9] | 36.8 [27.2 to 47.4]
  FU Year 2 | 30.1 [21.0 to 40.5] | 38.2 [28.1 to 49.1] | 33.0 [24.2 to 42.8] | 48.4 [38.0 to 58.9]
  FU Year 3 | 41.9 [31.8 to 52.6] | 46.1 [35.4 to 57.0] | 38.7 [29.4 to 48.6] | 53.7 [43.2 to 64.0]
  FU Year 4 | 46.2 [35.8 to 56.9] | 49.4 [38.7 to 60.2] | 49.1 [39.2 to 59.0] | 53.7 [43.2 to 64.0]
  FU Year 5 | 50.5 [40.0 to 61.1] | 49.4 [38.7 to 60.2] | 50.0 [40.1 to 59.9] | 51.6 [41.1 to 62.0]

3. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroconversion.
Description: HBsAg seroconversion was defined as the absence of HBsAg (a negative result for HBsAg) and the presence of anti-HBs (a positive result for anti-HBs). Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 0.0 [0.0 to 3.9] | 1.1 [0.0 to 6.1] | 1.9 [0.2 to 6.6] | 3.2 [0.7 to 9.0]
  FU Year 1 | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 4.1] | 0.9 [0.0 to 5.1] | 1.1 [0.0 to 5.7]
  FU Year 2 | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 4.1] | 0.9 [0.0 to 5.1] | 3.2 [0.7 to 9.0]
  FU Year 3 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 0.9 [0.0 to 5.1] | 3.2 [0.7 to 9.0]
  FU Year 4 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 0.9 [0.0 to 5.1] | 2.1 [0.3 to 7.4]
  FU Year 5 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 1.9 [0.2 to 6.6] | 2.1 [0.3 to 7.4]

4. Secondary Outcome: Percentage of Participants With Presence of Anti-Hepatitis B Envelope Antigen (HBe).
Description: The presence of anti-HBe is defined as antibody produced against e antigen in HBeAg. Seroconversion from e antigen to e antibody (anti-HBe) is a predictor of long-term clearance of hepatitis B virus (HBV) in participants undergoing antiviral therapy and indicates lower levels of HBV, and therefore lower infectivity. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 23.7 [15.5 to 33.6] | 27.0 [18.1 to 37.4] | 29.2 [20.8 to 38.9] | 40.0 [30.1 to 50.6]
  FU Year 1 | 28.0 [19.1 to 38.2] | 42.7 [32.3 to 53.6] | 28.3 [20.0 to 37.9] | 38.9 [29.1 to 49.5]
  FU Year 2 | 31.2 [22.0 to 41.6] | 40.4 [30.2 to 51.4] | 33.0 [24.2 to 42.8] | 50.5 [40.1 to 60.9]
  FU Year 3 | 41.9 [31.8 to 52.6] | 42.7 [32.3 to 53.6] | 36.8 [27.6 to 46.7] | 55.8 [45.2 to 66.0]
  FU Year 4 | 37.6 [27.8 to 48.3] | 44.9 [34.4 to 55.9] | 41.5 [32.0 to 51.5] | 52.6 [42.1 to 63.0]
  FU Year 5 | 43.0 [32.8 to 53.7] | 48.3 [37.6 to 59.2] | 42.5 [32.9 to 52.4] | 50.5 [40.1 to 60.9]

5. Secondary Outcome: Percentage of Participants With Presence of Anti-HBs
Description: The presence of anti-HBs is defined as antibody produced against HBsAg.It is generally interpreted as indicating recovery and immunity from HBV infection. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 4.3 [1.2 to 10.6] | 2.2 [0.3 to 7.9] | 11.3 [6.0 to 18.9] | 9.5 [4.4 to 17.2]
  FU Year 1 | 6.5 [2.4 to 13.5] | 3.4 [0.7 to 9.5] | 7.5 [3.3 to 14.3] | 7.4 [3.0 to 14.6]
  FU Year 2 | 5.4 [1.8 to 12.1] | 10.1 [4.7 to 18.3] | 6.6 [2.7 to 13.1] | 6.3 [2.4 to 13.2]
  FU Year 3 | 4.3 [1.2 to 10.6] | 4.5 [1.2 to 11.1] | 7.5 [3.3 to 14.3] | 5.3 [1.7 to 11.9]
  FU Year 4 | 4.3 [1.2 to 10.6] | 3.4 [0.7 to 9.5] | 4.7 [1.5 to 10.7] | 5.3 [1.7 to 11.9]
  FU Year 5 | 3.2 [0.7 to 9.1] | 4.5 [1.2 to 11.1] | 5.7 [2.1 to 11.9] | 5.3 [1.7 to 11.9]

6. Secondary Outcome: Percentage of Participants With Normalised Alanine Transaminase (ALT)
Description: Alanine Transaminase is an enzyme found mainly in liver and is measured to check if the liver is damaged or diseased. In case of liver damage or disease, the liver releases ALT into the blood stream and the ALT levels increase. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 28.0 [19.1 to 38.2] | 27.0 [18.1 to 37.4] | 38.7 [29.4 to 48.6] | 49.5 [39.1 to 59.9]
  FU Year 1 | 45.2 [34.8 to 55.8] | 44.9 [34.4 to 55.9] | 49.1 [39.2 to 59.0] | 50.5 [40.1 to 60.9]
  FU Year 2 | 58.1 [47.4 to 68.2] | 60.7 [49.7 to 70.9] | 55.7 [45.7 to 65.3] | 65.3 [54.8 to 74.7]
  FU Year 3 | 66.7 [56.1 to 76.1] | 70.8 [60.2 to 79.9] | 54.7 [44.8 to 64.4] | 66.3 [55.9 to 75.7]
  FU Year 4 | 67.7 [57.3 to 77.1] | 64.0 [53.2 to 73.9] | 62.3 [52.3 to 71.5] | 63.2 [52.6 to 72.8]
  FU Year 5 | 69.9 [59.5 to 79.0] | 67.4 [56.7 to 77.0] | 56.6 [46.6 to 66.2] | 63.2 [52.6 to 72.8]

7. Primary Outcome: Percentage of Participants With HBsAg Loss
Description: HBsAg loss is defined as the absence of HBsAg (i.e. a negative result for HBsAg). Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage
  EOT | 0.0 [0.0 to 3.9] | 1.1 [0.0 to 6.1] | 1.9 [0.2 to 6.6] | 3.2 [0.7 to 9.0]
  FU Year 1 | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 4.1] | 0.9 [0.0 to 5.1] | 1.1 [0.0 to 5.7]
  FU Year 2 | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 4.1] | 1.9 [0.2 to 6.6] | 3.2 [0.7 to 9.0]
  FU Year 3 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 1.9 [0.2 to 6.6] | 3.2 [0.7 to 9.0]
  FU Year 4 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 2.8 [0.6 to 8.0] | 2.1 [0.3 to 7.4]
  FU Year 5 | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 4.1] | 2.8 [0.6 to 8.0] | 2.1 [0.3 to 7.4]

8. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) Suppression < 20,000 International Unit/Milliliter (IU/mL).
Description: The percentage of participants with HBV-DNA suppression < 20,000 IU/mL. HBV DNA is the genetic material that carries the blueprint of the virus. The measure of HBV DNA in blood indicates how rapidly the virus is replicating in liver. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 22.6 [14.6 to 32.4] | 33.7 [24.0 to 44.5] | 34.0 [25.0 to 43.8] | 50.5 [40.1 to 60.9]
  FU Year 1 | 33.3 [23.9 to 43.9] | 31.5 [22.0 to 42.2] | 45.3 [35.6 to 55.2] | 40.0 [30.1 to 50.6]
  FU Year 2 | 57.0 [46.3 to 67.2] | 50.6 [39.8 to 61.3] | 58.5 [48.5 to 68.0] | 54.7 [44.2 to 65.0]
  FU Year 3 | 67.7 [57.3 to 77.1] | 61.8 [50.9 to 71.9] | 61.3 [51.4 to 70.6] | 64.2 [53.7 to 73.8]
  FU Year 4 | 69.9 [59.5 to 79.0] | 68.5 [57.8 to 78.0] | 68.9 [59.1 to 77.5] | 64.2 [53.7 to 73.8]
  FU Year 5 | 67.7 [57.3 to 77.1] | 70.8 [60.2 to 79.9] | 67.0 [57.2 to 75.8] | 63.2 [52.6 to 72.8]

9. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) Suppression < 2,000 International Unit/Milliliter (IU/mL)
Description: The percentage of participants with HBV-DNA suppression < 2,000 IU/mL. HBV DNA is the genetic material that carries the blueprint of the virus. The measure of HBV DNA in blood indicates how rapidly the virus is replicating in liver. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 15.1 [8.5 to 24.0] | 21.3 [13.4 to 31.3] | 27.4 [19.1 to 36.9] | 45.3 [35.0 to 55.8]
  FU Year 1 | 20.4 [12.8 to 30.1] | 23.6 [15.2 to 33.8] | 39.6 [30.3 to 49.6] | 31.6 [22.4 to 41.9]
  FU Year 2 | 45.2 [34.8 to 55.8] | 39.3 [29.1 to 50.3] | 50.0 [40.1 to 59.9] | 45.3 [35.0 to 55.8]
  FU Year 3 | 52.7 [42.1 to 63.1] | 52.8 [41.9 to 63.5] | 52.8 [42.9 to 62.6] | 52.6 [42.1 to 63.0]
  FU Year 4 | 59.1 [48.5 to 69.2] | 56.2 [45.3 to 66.7] | 63.2 [53.3 to 72.4] | 54.7 [44.2 to 65.0]
  FU Year 5 | 59.1 [48.5 to 69.2] | 61.8 [50.9 to 71.9] | 60.4 [50.4 to 69.7] | 57.9 [47.3 to 68.0]

10. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) Suppression < 80 International Unit/Milliliter (IU/mL)
Description: The percentage of participants with HBV-DNA suppression < 80 IU/mL. HBV DNA is the genetic material that carries the blueprint of the virus. The measure of HBV DNA in blood indicates how rapidly the virus is replicating in liver. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Percentage of participants
  EOT | 5.4 [1.8 to 12.1] | 12.4 [6.3 to 21.0] | 16.0 [9.6 to 24.4] | 32.6 [23.4 to 43.0]
  FU Year 1 | 12.9 [6.8 to 21.5] | 7.9 [3.2 to 15.5] | 17.9 [11.2 to 26.6] | 14.7 [8.3 to 23.5]
  FU Year 2 | 28.0 [19.1 to 38.2] | 23.6 [15.2 to 33.8] | 36.8 [27.6 to 46.7] | 29.5 [20.6 to 39.7]
  FU Year 3 | 39.8 [29.8 to 50.5] | 30.3 [21.0 to 41.0] | 34.9 [25.9 to 44.8] | 38.9 [29.1 to 49.5]
  FU Year 4 | 47.3 [36.9 to 57.9] | 38.2 [28.1 to 49.1] | 46.2 [36.5 to 56.2] | 40.0 [30.1 to 50.6]
  FU Year 5 | 39.8 [29.8 to 50.5] | 40.4 [30.2 to 51.4] | 42.5 [32.9 to 52.4] | 38.9 [29.1 to 49.5]

11. Secondary Outcome: Quantitative HBsAg
Description: Quantitative HBsAg assay is a diagnostic test for assessing the amount of the HBsAg in chronic Hepatitis B participants. Missing values were counted as non-response.
Time Frame: Annually, for up to 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
log10 IU/mL
  EOT (n= 89, 86, 102, 91) | 3.541 (0.9523) | 3.371 (1.1570) | 3.322 (1.0875) | 2.949 (1.3170)
  FU Year 1 (n= 87, 85, 93, 86) | 3.495 (0.9314) | 3.484 (0.8102) | 3.379 (0.9076) | 3.453 (0.9282)
  FU Year 2 (n= 86, 86, 96, 90) | 3.478 (0.9263) | 3.441 (0.7682) | 3.381 (0.8898) | 3.318 (1.0139)
  FU Year 3 (n= 83, 82, 91, 85) | 3.479 (0.9008) | 3.393 (0.7095) | 3.339 (0.8870) | 3.178 (1.0561)
  FU Year 4 (n= 81, 79, 89, 80) | 3.456 (0.9418) | 3.350 (0.8172) | 3.240 (0.9143) | 3.135 (0.9906)
  FU Year 5 (n= 81, 79, 83, 74) | 3.391 (0.8555) | 3.305 (0.8206) | 3.201 (0.9099) | 2.932 (1.1391)

12. Secondary Outcome: Number of Participants Who Received Treatment With Antiviral, Immunomodulatory, Anti-inflammatory or Herbal/Botanical/Other Treatments for Chronic Hepatitis B
Description: Participants who required additional treatments specifically to treat CHB, associated laboratory test abnormalities and associated symptoms in this long-term observation in the study were reported. Receipt of such treatment did not require participant withdrawal from further participation.
Time Frame: Up to 5-year FU period
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Group A: Participants received 90 mcg PEG-IFN SC once a week for 24 weeks in Study WV19432 and entered FU Study MV22430.
- Group B: Participants received 180 mcg PEG-IFN SC once a week for 24 weeks in Study WV19432 and entered FU Study MV22430.
- Group C: Participants received 90 mcg PEG-IFN SC once a week for 48 weeks in Study WV19432 and entered FU Study MV22430.
- Group D: Participants received 180 mcg PEG-IFN SC once a week for 48 weeks in Study WV19432 and entered FU Study MV22430.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 93 | 89 | 106 | 95
Participants
  Nucleoside/nucleotide analogues | 49 | 40 | 51 | 36
  Antiviral agents | 9 | 7 | 18 | 9
  Cytokines | 2 | 8 | 9 | 9
  Botanicals | 4 | 6 | 4 | 9
  Miscellaneous gastrointestinal agents | 5 | 3 | 4 | 7
  Miscellaneous drugs | 1 | 1 | 2 | 1
  Supplements | 2 | 1 | 1 | 0
  Pharmaceutic aids | 1 | 1 | 1 | 0
  Immunomodulators | 0 | 2 | 0 | 0
  Blood products | 0 | 1 | 0 | 0
  Chelating agents | 0 | 1 | 0 | 0
  Clotting factors and haemostatics | 0 | 1 | 0 | 0
  Prostaglandins | 0 | 1 | 0 | 0
  Vaccines, toxoids and serologic agents | 0 | 1 | 0 | 0
  Vitamins and minerals | 1 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Events Related to Chronic Hepatitis B (CHB)
Description: Clinically significant events were defined as one or more of the following: Hepatocellular carcinoma, hepatic decompensation, CHB-related death, hepatic transplant, marked elevation of serum ALT of >10 x upper limit of normal (ULN).
Time Frame: Up to 5-year FU period
Population: The safety analysis population included participants who had received at least one dose of study medication in Study WV19432, had at least one visit in study MV22430. Analysis was performed as per the treatment received and not the randomized treatment. Four participants in the safety population switched treatment groups.
Measure: Number; unit: Participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Participants
  Elevated ALT >10 x ULN (Yes) | 3 | 5 | 9 | 5
  Elevated ALT >10 x ULN (No) | 89 | 83 | 97 | 90
  Elevated ALT >10 x ULN (Missing) | 1 | 1 | 0 | 0
  Hepatic Decompensation (Yes) | 2 | 0 | 1 | 1
  Hepatic Decompensation (No) | 88 | 87 | 105 | 94
  Hepatic Decompensation (Missing) | 3 | 2 | 0 | 0
  Hepatocellular Carcinoma (Yes) | 1 | 0 | 3 | 0
  Hepatocellular Carcinoma (No) | 20 | 22 | 22 | 21
  Hepatocellular Carcinoma (No assessment performed) | 71 | 66 | 81 | 74
  Hepatocellular Carcinoma (Missing) | 1 | 1 | 0 | 0
  Hepatic Transplant (No) | 92 | 88 | 106 | 95
  Hepatic Transplant (Missing) | 1 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Marked abnormality of laboratory parameters is defined as the value which is outside the defined reference range of that respective parameter. Roche's following reference ranges for laboratory test parameters were used for the analysis: Hemoglobin (reference range: 110-200 grams/liter[g/L]), White blood cells (WBC) (3.0-18.0 ^10^9/L), Platelets (100-550 ^10^9/L), Neutrophils (1.50-9.25 ^10^9/L), Prothrombin time (PT) Normal ratio (n.d.-2.00), Alkaline phosphatase (0-220 units/liter [U/L]), Alanine aminotransferase (0-110 U/L), Aspartate transaminase (0-80 U/L), Total bilirubin (0-34 micromole/liter [umol/L]), Gamma-glutamyl transpeptidase (GGT) (0-190 U/L), Blood urea nitrogen (BUN) (0.0-14.3 millimole/liter [mmol/L]), Creatinine (0-154 umol/L), Total Protein (55-87 g/L), Albumin (30.0-n.d. g/L), Potassium (2.9-5.8 mmol/L), Sodium (130-150 mmol/L), Calcium (2.00-2.90 mmol/L), Uric acid (0-600 umol/L). It includes marked abnormalities observed during Study WV19432 and FU study MV22430
Time Frame: Up to 5-year FU period
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Number analyzed (Participants) | 93 | 89 | 106 | 95
Participants
  Alanine transaminase (High) | 66 | 67 | 74 | 56
  Aspartate transaminase (High) | 60 | 60 | 60 | 51
  Albumin (Low) | 1 | 2 | 1 | 0
  Alkaline phosphatase (High) | 0 | 2 | 1 | 1
  BUN (High) | 0 | 0 | 1 | 0
  Calcium (High) | 0 | 0 | 1 | 2
  Calcium (Low) | 5 | 5 | 15 | 7
  Creatinine (High) | 0 | 0 | 1 | 0
  GGT (High) | 3 | 5 | 7 | 7
  Hemoglobin (Low) | 5 | 6 | 1 | 13
  Neutrophils (High) | 3 | 2 | 2 | 2
  Neutrophils (Low) | 53 | 57 | 79 | 77
  PT normalized ratio (High) | 0 | 1 | 0 | 0
  Platelets (Low) | 14 | 23 | 28 | 41
  Potassium (High) | 2 | 1 | 4 | 2
  Potassium (Low) | 1 | 0 | 0 | 1
  Prothrombin time (High) | 0 | 1 | 1 | 0
  Sodium (High) | 3 | 0 | 1 | 0
  Sodium (Low) | 0 | 0 | 1 | 0
  Total bilirubin (High) | 2 | 4 | 8 | 3
  Total protein (High) | 3 | 1 | 5 | 6
  Total Protein (Low) | 1 | 0 | 1 | 0
  Uric acid (High) | 1 | 1 | 2 | 1
  White blood cell (Low) | 27 | 34 | 52 | 65

ADVERSE EVENTS:
Time Frame: 5-year FU period
Description: Serious adverse events and non-serious adverse events are reported in safety analysis set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | PEG-IFN 90mcg 24 Wks | PEG-IFN 180mcg 24 Wks | PEG-IFN 90mcg 48 Wks | PEG-IFN 180mcg 48 Wks
Serious Adverse Events (participants affected / at risk) | 5/93 | 4/89 | 10/106 | 6/95
Other Adverse Events (participants affected / at risk) | 8/93 | 8/89 | 8/106 | 12/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN 90mcg 24 Wks (N=93) | PEG-IFN 180mcg 24 Wks (N=89) | PEG-IFN 90mcg 48 Wks (N=106) | PEG-IFN 180mcg 48 Wks (N=95)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN 90mcg 24 Wks (N=93) | PEG-IFN 180mcg 24 Wks (N=89) | PEG-IFN 90mcg 48 Wks (N=106) | PEG-IFN 180mcg 48 Wks (N=95)
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 4 | 7
Alanine aminotransferase increased (Investigations) | 3 | 2 | 4 | 5

LIMITATIONS AND CAVEATS:
Of the responders at FU Year 5, the proportion of patients who were receiving additional anti-HBV treatment after FU Week 24 varied between groups.

The frequency of missing values (counted as non-response) was unevenly distributed between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.